CLINICAL TRIAL: NCT00819390
Title: A Phase II, Double Blind, Randomized, Exploratory Study of Chloroquine for Reducing HIV-Associated Immune Activation
Brief Title: Chloroquine for Reducing Immune Activation in HIV- Infected Individuals
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACTG A5258; 1U01AI068636 (NIH)
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Results first posted 2014-09-05 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Chloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A: Chloroquine then Placebo for Off-ART Participants (Experimental): Participants received chloroquine treatment from Day 0 through the Week 12 study visit and then began chloroquine placebo treatment until the Week 24 study visit.
  Interventions: Drug: Chloroquine; Drug: Placebo
- B: Placebo then Chloroquine for Off-ART Participants (Experimental): Participants received chloroquine placebo treatment from Day 0 through the Week 12 study visit and then began chloroquine treatment until the Week 24 study visit.
  Interventions: Drug: Chloroquine; Drug: Placebo
- C: Chloroquine then Placebo for On-ART Participants (Experimental): Participants received chloroquine treatment from Day 0 through the Week 12 study visit and then began chloroquine placebo treatment until the Week 24 study visit.
  Interventions: Drug: Chloroquine; Drug: Placebo
- D: Placebo then Chloroquine for On-ART Participants (Experimental): Participants received chloroquine placebo treatment from Day 0 through the Week 12 study visit and then began chloroquine treatment until the Week 24 study visit.
  Interventions: Drug: Chloroquine; Drug: Placebo

INTERVENTIONS:
Drug: Chloroquine — Taken orally, once daily, at a dose of 250 mg for 12 weeks.
Drug: Placebo — Taken orally, once daily for 12 weeks.

SUMMARY:
HIV is characterized by frequent immune system activation. Early in the course of infection the body establishes an immune activation "set point" related to the amount of HIV in the blood stream. This set point affects the rate of CD4 cell loss. Without CD4 cells, or with very low levels of CD4 cells, the body cannot fight off illness. This is known as immunodeficiency. If left untreated HIV can lead to extreme immunodeficiency and AIDS.

Evidence suggests that by decreasing the rate of immune system activation, immune deficiency progression could be prevented. The purpose of this study is to learn how well chloroquine can reduce the level of immune activation and to test the safety and tolerance of chloroquine in people infected with HIV.

DETAILED DESCRIPTION:
HIV is characterized by persistent immune system activation, and early in the course of infection the body establishes an immune activation "set point" related to the amount of HIV in the blood stream. This set point affects the rate of CD4 cell loss. Without CD4 cells, or with very low levels of CD4 cells, the body cannot fight off illness. This is known as immunodeficiency. If left untreated HIV can lead to extreme immunodeficiency and AIDS.

Immune system activation includes activating the CD8 cells. These cells attack body cells infected with viruses. Because of this, CD4 cells infected with HIV are frequently destroyed by CD8 cells. The purpose of this study is to learn how well chloroquine reduces the level of activation of CD8 cells in people infected with HIV. Increased activation of CD8 cells is thought to lead to a more severe path of disease in HIV infection.

The constant immune activation observed in HIV- infected patients has also been linked to higher levels of byproducts from certain naturally occurring bacteria found in the gut that are known to be immune stimulants. By decreasing the stimulation from these byproducts with chloroquine treatment, HIV disease may be slowed.

The purpose of this study was to learn how well chloroquine reduces the level of activation of CD8 cells and lowers the levels of bacteria byproducts in people infected with HIV, either off antiretroviral therapy (ART) (protocol version 1.0 dated December 17, 2008) or on-ART (protocol version 2.0 dated October 1, 2010). The off-ART (Arms A and B) and on-ART (Arms C and D) participants were enrolled during different time periods, and the study was designed to analyze the two study populations separately. This study also looked at how well chloroquine was tolerated and its safety in HIV- infected participants.

Off-ART participants in the study were randomized with equal probability to one of two treatment arms:

Arm A: Participants received 12 weeks of chloroquine treatment followed by 12 weeks of placebo

Arm B: Participants received 12 weeks of placebo followed by 12 weeks of chloroquine

On-ART participants in the study were randomized with equal probability to one of two treatment arms:

Arm C: Participants received 12 weeks of chloroquine treatment followed by 12 weeks of placebo

Arm D: Participants received 12 weeks of placebo followed by 12 weeks of chloroquine

Study treatment was given once a day for a full 24 weeks. There was an additional 4 weeks of follow-up for purposes of safety. After treatment has started, participants were asked to come to the clinic on Weeks 4, 10, 12, 16, 22, and 24. At each visit participants were given enough study treatment to last until the next visit. Each visit lasted between 30 and 60 minutes. At most visits, participants had a physical exam, answered questions about any medications they were taking and how they are feeling, and had blood drawn for safety to assess CD4/CD8 cell counts and viral load. Some additional blood were also stored for immunology testing. At some visits, participants were asked questions about their medication and medical history, had pupils dilated, had a hearing test, and had an electrocardiogram (EKG). Some visits required participants to arrive fasting. Pregnancy tests were also conducted if the participant is able to become pregnant or if pregnancy was suspected.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected
* Certain specified laboratory values obtained within 30 days prior to study entry. More information on this criterion can be found in the study protocol.
* Documentation that pre-entry specimen for the primary immune activation endpoint responses has been obtained
* Female participants of reproductive potential must have a negative pregnancy test performed within 24 hours prior to study entry
* If engaging in sexual activity, female participants must use adequate forms of contraception while receiving study treatment and for 4 weeks after stopping the treatment. More information on this criterion can be found in the study protocol.
* Ability and willingness to provide informed consent

Additional Inclusion Criteria for Off-ART Participants:

* No antiretroviral therapy (ART) for at least 6 months prior to study entry and not likely to start within the 6 months after study entry
* CD4 cell count greater than or equal to 400 cells/mm3 at screening, obtained within 30 days prior to study entry
* For participants with previous ART use, documentation or recall of nadir CD4 cell count greater than or equal to 200 cells/mm3
* HIV-1 RNA viral load greater than or equal to 1,000 copies/mL obtained within 30 days prior to study entry
* No history of CDC category C AIDS-related opportunistic infections
* Karnofsky performance score greater than or equal to 70 within 30 days prior to study entry

Additional Inclusion Criteria for On-ART Participants:

* Receiving ART, defined as a regimen that includes three or more antiretroviral medications, for at least 24 months prior to study entry
* Required documentation that all HIV-1 viral loads (at least two) were below 400 copies/mL. More information on this criterion can be found in the study protocol.
* Screening HIV-1 RNA <200 copies/mL within 30 days prior to study entry. More information on this criterion can be found in the study protocol.
* CD4 cell count <350 cells/mm3 at screening, obtained within 30 days prior to study entry

Exclusion Criteria:

* Continuous use of certain specified medication for more than 3 days within 30 days prior to study entry. More information on this criterion can be found in the study protocol.
* Use of chloroquine or hydroxychloroquine within 3 months prior to study entry
* Known history of hypersensitivity to 4-aminoquinoline compounds (such as chloroquine or hydroxychloroquine)
* Active drug or alcohol use or dependence that, in the opinion of the investigator would interfere with adherence to study requirements
* Serious illness requiring systemic treatment and/or hospitalization within 30 days prior to study entry
* Renal insufficiency, defined as serum creatinine greater than 1.5 mg/dL, within 30 days prior to study entry
* History of retinal disease (i.e. confirmed retinopathy by ophthalmologic examination)
* History of neoplasm, within 5 years prior to study entry, other than treated in situ carcinoma or basal-cell or localized squamous cell carcinoma of the skin
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency at screening
* History of porphyria
* History of psoriasis
* History of cirrhosis
* History of seizure disorder
* History of tinnitus (ear and/or head noise lasting more than 5 minutes that occurs more often than once per week) or history of sudden hearing loss
* History of myopathy
* History of cardiac conduction abnormality or cardiomyopathy. More information on this criterion can be found in the study protocol.

Additional Exclusion Criteria for On-ART Participants:

- Plans to change ART regimen with the 6 months after study entry (change in ART regimen is only permitted if due to toxicity)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-03; Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M Jacobson, MD, Study Chair — Drexel University College of Medicine
Locations (15):
- United States (15):
  - Alabama Therapeutics CRS (5801), Birmingham, Alabama
  - Ucsd, Avrc Crs (701), San Diego, California
  - University of Colorado Hospital CRS (6101), Aurora, Colorado
  - Georgetown University CRS (GU CRS) (1008), Washington D.C., District of Columbia
  - Johns Hopkins Adult AIDS CRS (201), Baltimore, Maryland
  - Massachusetts General Hospital ACTG CRS (101), Boston, Massachusetts
  - Washington University CRS (2101), St Louis, Missouri
  - Cornell CRS (7804), New York, New York
  - Unc Aids Crs (3201), Chapel Hill, North Carolina
  - Univ. of Cincinnati CRS (2401), Cincinnati, Ohio
  - Case CRS (2501), Cleveland, Ohio
  - MetroHealth CRS (2503), Cleveland, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS (6201), Philadelphia, Pennsylvania
  - Pittsburgh CRS (1001), Pittsburgh, Pennsylvania
  - Vanderbilt Therapeutics CRS (3652), Nashville, Tennessee

REFERENCES:
- [Background] Neely M, Kalyesubula I, Bagenda D, Myers C, Olness K. Effect of chloroquine on human immunodeficiency virus (HIV) vertical transmission. Afr Health Sci. 2003 Aug;3(2):61-7. PMID 12913796
- [Background] Savarino A, Boelaert JR, Cassone A, Majori G, Cauda R. Effects of chloroquine on viral infections: an old drug against today's diseases? Lancet Infect Dis. 2003 Nov;3(11):722-7. doi: 10.1016/s1473-3099(03)00806-5. PMID 14592603
- [Background] Semrau K, Kuhn L, Kasonde P, Sinkala M, Kankasa C, Shutes E, Vwalika C, Ghosh M, Aldrovandi G, Thea DM. Impact of chloroquine on viral load in breast milk. Trop Med Int Health. 2006 Jun;11(6):800-3. doi: 10.1111/j.1365-3156.2006.01645.x. PMID 16772000
- [Derived] Jacobson JM, Bosinger SE, Kang M, Belaunzaran-Zamudio P, Matining RM, Wilson CC, Flexner C, Clagett B, Plants J, Read S, Purdue L, Myers L, Boone L, Tebas P, Kumar P, Clifford D, Douek D, Silvestri G, Landay AL, Lederman MM. The Effect of Chloroquine on Immune Activation and Interferon Signatures Associated with HIV-1. AIDS Res Hum Retroviruses. 2016 Jul;32(7):636-47. doi: 10.1089/AID.2015.0336. Epub 2016 Apr 19. PMID 26935044

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Version 1.0 of the study enrolled off antiretroviral therapy (ART) participants only. Off-ART participants were enrolled from March 2009 to July 2010.
  On-ART participants were allowed to enroll in Version 2.0 of the study. On-ART participants were enrolled from December 2010 to November 2012.
Pre-assignment Details: Analysis of data from off-ART and on-ART participants was done separately. The study analyses did not utilize the cross-over design, and the primary analysis consists of comparison between the chloroquine and placebo arms after the first 12 weeks on study in each off-ART and on-ART study populations.
Period: Overall Study
Arm/Group | A: Chloroquine Then Placebo for Off-ART Participants | B: Placebo Then Chloroquine for Off-ART Participants | C: Chloroquine Then Placebo for On-ART Participants | D: Placebo Then Chloroquine for On-ART Participants
Started | 16 | 17 | 18 | 19
Completed | 13 | 16 | 17 | 19
Not Completed | 3 | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Results are for all participants, off-ART and on-ART, who enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | A: Chloroquine Then Placebo for Off-ART Participants | B: Placebo Then Chloroquine for Off-ART Participants | C: Chloroquine Then Placebo for On-ART Participants | D: Placebo Then Chloroquine for On-ART Participants | Total
Number analyzed (Participants) | 16 | 17 | 18 | 19 | 70
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 35 [29 to 43] | 39 [35 to 44] | 50 [48 to 55] | 49 [41 to 56] | 46 [36 to 50]
Age, Customized [Number; unit: participants]
  18-29 years | 5 | 2 | 1 | 0 | 8
  30-39 years | 5 | 7 | 1 | 3 | 16
  40-49 years | 5 | 8 | 5 | 7 | 25
  50-59 years | 1 | 0 | 10 | 7 | 18
  60-69 years | 0 | 0 | 0 | 2 | 2
  70-79 years | 0 | 0 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 2 | 7
  Male | 14 | 15 | 17 | 17 | 63
Region of Enrollment [Number; unit: participants]
  United States | 16 | 17 | 18 | 19 | 70

OUTCOME MEASURES:

1. Primary Outcome: Change in Percent CD8 HLA-DR+/CD38+ From Baseline to Week 12
Description: The baseline percent CD8 HLA-DR+/CD38+ (mean of pre-entry and entry percent CD8 HLA-DR+/CD38+) was subtracted from the mean of week 10 and week 12 percent CD8 HLA-DR+/CD38+.
Time Frame: At pre-entry, entry, weeks 10 and 12
Population: Analysis used a modified as-treated approach, limited to participants with assay data at baseline and weeks 10 or 12, and with no break in study treatment for >=14 days. Off-ART analysis excluded participants who started ART. On-ART analysis excluded participants who stopped ART or had virologic rebound (confirmed HIV-1 RNA>1000 copies/mL).
Measure: Median (Inter-Quartile Range); unit: percent of CD8 expressing HLA-DR+/CD38+
Arm/Group | A: Chloroquine Then Placebo for Off-ART Participants | B: Placebo Then Chloroquine for Off-ART Participants | C: Chloroquine Then Placebo for On-ART Participants | D: Placebo Then Chloroquine for On-ART Participants
Number analyzed (Participants) | 15 | 16 | 16 | 19
percent of CD8 expressing HLA-DR+/CD38+ | -2.0 [-10.0 to 9.0] | -0.5 [-2.3 to 2.8] | -3.1 [-4.3 to 0.4] | -1.2 [-3.3 to 1.4]
Statistical Analysis 1: Comparison: A: Chloroquine Then Placebo for Off-ART Participants vs B: Placebo Then Chloroquine for Off-ART Participants; Null hypothesis: There is no difference between the two arms/groups with respect to change in percent CD8 HLA-DR+/CD38+ from baseline to week 12; Test type: Superiority or Other; p = 0.428, Wilcoxon (Mann-Whitney) — The p-value is not adjusted for multiple comparisons. The a priori threshold for statistical significance used for the two-sided test was 0.05; No other adjustments
Statistical Analysis 2: Comparison: C: Chloroquine Then Placebo for On-ART Participants vs D: Placebo Then Chloroquine for On-ART Participants; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.247, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]; No other adjustments

2. Secondary Outcome: Change in Percent CD8 HLA-DR+/CD38+ From Start to End of the 12-week Chloroquine Treatment Period
Description: For Arm A: Chloroquine then Placebo for off-ART participants and Arm C: Chloroquine then Placebo for on-ART participants, the baseline percent CD8 HLA-DR+/CD38+ (mean of pre-entry and entry percent CD8 HLA-DR+/CD38+) was subtracted from the mean of week 10 and week 12 percent CD8 HLA-DR+/CD38+. For Arm B: Placebo then Chloroquine for off-ART participants and Arm D: Placebo then Chloroquine for on-ART participants, the mean of week 10 and week 12 percent CD8 HLA-DR+/CD38+ was subtracted from the mean of week 22 and week 24 percent CD8 HLA-DR+/CD38+.
Time Frame: For Arms A and C: Pre-entry, entry, weeks 10 and 12. For Arms B and D: Weeks 10, 12, 22 and 24
Population: Analysis used a modified as-treated approach, limited to participants with assay data at the required time points, and with no break in study treatment for >=14 days. Off-ART analysis excluded participants who started ART. On-ART analysis excluded participants who stopped ART or had virologic rebound (confirmed HIV-1 RNA>1000 copies/mL).
Measure: Median (Inter-Quartile Range); unit: percent of CD8 expressing HLA-DR+/CD38+
Arm/Group | A: Chloroquine Then Placebo for Off-ART Participants | B: Placebo Then Chloroquine for Off-ART Participants | C: Chloroquine Then Placebo for On-ART Participants | D: Placebo Then Chloroquine for On-ART Participants
Number analyzed (Participants) | 15 | 13 | 16 | 18
percent of CD8 expressing HLA-DR+/CD38+ | -2.0 [-10.0 to 9.0] | 1.5 [-2.5 to 7.0] | -3.1 [-4.3 to 0.4] | -2.9 [-4.7 to -0.4]

3. Secondary Outcome: Change in Percent CD8 HLA-DR+/CD38+ From Week 12 to Week 24
Description: The mean of week 10 and week 12 percent CD8 HLA-DR+/CD38+ is subtracted from the mean of the week 22 and week 24 percent CD8 HLA-DR+/CD38+
Time Frame: At Weeks 10, 12, 22 and 24
Population: Analysis used a modified as-treated approach, limited to participants with assay data at weeks 10 or 12, and 22 or 24, and with no break in study treatment for >=14 days. Off-ART analysis excluded participants who started ART. On-ART analysis excluded participants who stopped ART or had virologic rebound (confirmed HIV-1 RNA>1000 copies/mL).
Measure: Median (Inter-Quartile Range); unit: percent of CD8 expressing HLA-DR+/CD38+
Arm/Group | A: Chloroquine Then Placebo for Off-ART Participants | B: Placebo Then Chloroquine for Off-ART Participants | C: Chloroquine Then Placebo for On-ART Participants | D: Placebo Then Chloroquine for On-ART Participants
Number analyzed (Participants) | 12 | 13 | 13 | 18
percent of CD8 expressing HLA-DR+/CD38+ | 5.5 [2.0 to 13.8] | 1.5 [-2.5 to 7.0] | -0.1 [-3.6 to 2.7] | -2.9 [-4.7 to -0.4]

4. Secondary Outcome: Change in Percent CD8 HLA-DR+/CD38+ From Baseline to Week 24 in Arm A and Arm C
Description: The baseline percent CD8 HLA-DR+/CD38+ (mean of pre-entry and entry percent CD8 HLA-DR+/CD38+) was subtracted from the mean of week 22 and week 24 percent CD8 HLA-DR+/CD38+.
Time Frame: At Pre-entry, entry, Weeks 22 and 24
Population: Analysis used a modified as-treated approach, limited to participants with assay data at baseline and weeks 22 or 24, and with no break in study treatment for >=14 days. Off-ART analysis excluded participants who started ART. On-ART analysis excluded participants who stopped ART or had virologic rebound (confirmed HIV-1 RNA>1000 copies/mL).
Measure: Median (Inter-Quartile Range); unit: percent of CD8 expressing HLA-DR+/CD38+
Arm/Group | A: Chloroquine Then Placebo for Off-ART Participants | C: Chloroquine Then Placebo for On-ART Participants
Number analyzed (Participants) | 12 | 13
percent of CD8 expressing HLA-DR+/CD38+ | 10.8 [0 to 14.8] | -2.4 [-4.5 to 0]

5. Secondary Outcome: Change in Total CD4 T Cell Count From Baseline to Week 12
Description: Baseline CD4 count (mean of pre-entry and entry CD4 count) is subtracted from the mean of week 10 and week 12 CD4 count
Time Frame: At pre-entry, entry, weeks 10 and 12
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | A: Chloroquine Then Placebo for Off-ART Participants | B: Placebo Then Chloroquine for Off-ART Participants | C: Chloroquine Then Placebo for On-ART Participants | D: Placebo Then Chloroquine for On-ART Participants
Number analyzed (Participants) | 15 | 16 | 16 | 19
cells/mm^3 | -27 [-150 to 4] | -11 [-38 to 71] | -6 [-21 to 10] | 7 [-17 to 23]

6. Secondary Outcome: Number of Participants With Events Grade 3 or Higher
Description: Events included signs and symptoms, laboratory abnormalities and/or clinical events grade 3 or higher which were described by site clinician blinded to the treatment arm as definitely or possibly related to the study treatment.
Time Frame: From start of study treatment to study completion at week 28
Population: Analysis is based on all enrolled participants, off-ART and on-ART, who received study treatment.
Measure: Number; unit: participants
Arm/Group | A: Chloroquine Then Placebo for Off-ART Participants | B: Placebo Then Chloroquine for Off-ART Participants | C: Chloroquine Then Placebo for On-ART Participants | D: Placebo Then Chloroquine for On-ART Participants
Number analyzed (Participants) | 16 | 17 | 18 | 19
participants | 0 | 1 | 1 | 0

7. Secondary Outcome: HIV-1 RNA Copies/mL at Study Entry for Off-ART Participants
Description: Results reported are for HIV-1 RNA (copies/mL) at study entry for off-ART participants.
Time Frame: At Entry
Population: Analysis is based on all off-ART participants with HIV-1 RNA data at entry.
Measure: Median (Inter-Quartile Range); unit: log10 copies/mL
Arm/Group | A: Chloroquine Then Placebo for Off-ART Participants | B: Placebo Then Chloroquine for Off-ART Participants
Number analyzed (Participants) | 16 | 17
log10 copies/mL | 4.48 [4.02 to 4.74] | 4.42 [4.03 to 4.83]

8. Secondary Outcome: HIV-1 RNA Copies/mL at Weeks 12 and 24 for Off-ART Participants
Description: Results reported are for HIV-1 RNA (copies/mL) at week 12 and week 24 for off-ART participants.
Time Frame: At weeks 12 and 24
Population: Analysis is based on all off-ART participants with HIV-1 RNA data at week 12 and week 24.
Measure: Median (Inter-Quartile Range); unit: log10 copies/mL
Arm/Group | A: Chloroquine Then Placebo for Off-ART Participants | B: Placebo Then Chloroquine for Off-ART Participants
Number analyzed (Participants) | 14 | 16
log10 copies/mL
  Week 12 | 4.68 [4.46 to 4.79] | 4.28 [4.08 to 4.60]
  Week 24 | 4.69 [4.31 to 4.90] | 4.61 [4.45 to 4.87]

9. Secondary Outcome: HIV-1 RNA Copies/mL at Study Entry for On-ART Participants
Description: Results reported are for HIV-1 RNA at study entry for on-ART participants.
Time Frame: At Entry
Population: Analysis is based on all on-ART participants with HIV-1 RNA data at entry.
Measure: Number; unit: participants
Arm/Group | C: Chloroquine Then Placebo for On-ART Participants | D: Placebo Then Chloroquine for On-ART Participants
Number analyzed (Participants) | 18 | 19
participants
  at or below lower limit of quantitation | 16 | 17
  above lower limit of quantitation | 2 | 2

10. Secondary Outcome: HIV-1 RNA Copies/mL at Week 12 for On-ART Participants
Description: Results reported are for HIV-1 RNA at week 12 for on-ART participants.
Time Frame: At week 12
Population: Analysis is based on all on-ART participants with HIV-1 RNA data at week 12.
Measure: Number; unit: participants
Arm/Group | C: Chloroquine Then Placebo for On-ART Participants | D: Placebo Then Chloroquine for On-ART Participants
Number analyzed (Participants) | 17 | 19
participants
  at or below lower limit of quantitation | 16 | 18
  above lower limit of quantitation | 1 | 1

11. Secondary Outcome: HIV-1 RNA Copies/mL at Week 24 for On-ART Participants
Description: Results reported are for HIV-1 RNA at week 24 for on-ART participants.
Time Frame: At week 24
Population: Analysis is based on all on-ART participants with HIV-1 RNA data at week 24.
Measure: Number; unit: participants
Arm/Group | C: Chloroquine Then Placebo for On-ART Participants | D: Placebo Then Chloroquine for On-ART Participants
Number analyzed (Participants) | 16 | 19
participants
  at or below lower limit of quantitation | 14 | 18
  above lower limit of quantitation | 2 | 1

12. Secondary Outcome: Percent CD8 CD38+ at Baseline
Description: Baseline CD8 CD38+ is computed as the mean of pre-entry and entry CD8 CD38+.
Time Frame: At pre-entry and entry
Population: Analysis is based on all participants with assay data at pre-entry or entry.
Measure: Median (Inter-Quartile Range); unit: percent of CD8 expressing CD38+
Arm/Group | A: Chloroquine Then Placebo for Off-ART Participants | B: Placebo Then Chloroquine for Off-ART Participants | C: Chloroquine Then Placebo for On-ART Participants | D: Placebo Then Chloroquine for On-ART Participants
Number analyzed (Participants) | 15 | 16 | 17 | 19
percent of CD8 expressing CD38+ | 71.0 [66.0 to 80.5] | 77.0 [71.5 to 88.3] | 50.8 [40.1 to 65.6] | 49.9 [37.8 to 63.5]

13. Secondary Outcome: Percent CD8 CD38+ at Week 12
Description: Results reported are the week 12 percentage of CD8 expressing CD38+.
Time Frame: At Week 12
Population: Analysis is based on all participants with assay data at week 12.
Measure: Median (Inter-Quartile Range); unit: percent of CD8 expressing CD38+
Arm/Group | A: Chloroquine Then Placebo for Off-ART Participants | B: Placebo Then Chloroquine for Off-ART Participants | C: Chloroquine Then Placebo for On-ART Participants | D: Placebo Then Chloroquine for On-ART Participants
Number analyzed (Participants) | 14 | 16 | 16 | 19
percent of CD8 expressing CD38+ | 71.5 [67.0 to 83.0] | 79.5 [69.0 to 88.5] | 50.9 [37.2 to 63.6] | 51.9 [38.7 to 63.0]

14. Secondary Outcome: Percent CD8 CD38+ at Week 24
Description: Results reported are the week 24 percentage of CD8 expressing CD38+.
Time Frame: At Week 24
Population: Analysis is based on all participants with assay data at week 24.
Measure: Median (Inter-Quartile Range); unit: percent of CD8 expressing CD38+
Arm/Group | A: Chloroquine Then Placebo for Off-ART Participants | B: Placebo Then Chloroquine for Off-ART Participants | C: Chloroquine Then Placebo for On-ART Participants | D: Placebo Then Chloroquine for On-ART Participants
Number analyzed (Participants) | 13 | 14 | 16 | 19
percent of CD8 expressing CD38+ | 78.0 [74.0 to 86.0] | 79.5 [69.0 to 89.0] | 50.6 [40.6 to 54.4] | 48.7 [38.2 to 64.9]

15. Secondary Outcome: Percent CD4 HLA-DR+/CD38+ at Baseline
Description: Baseline CD4 HLA-DR+/CD38+ is computed as the mean of pre-entry and entry CD4 HLA-DR+/CD38+.
Time Frame: At pre-entry and entry
Population: Analysis is based on all participants with assay data at pre-entry or entry.
Measure: Median (Inter-Quartile Range); unit: percent of CD4 expressing HLA-DR+/CD38+
Arm/Group | A: Chloroquine Then Placebo for Off-ART Participants | B: Placebo Then Chloroquine for Off-ART Participants | C: Chloroquine Then Placebo for On-ART Participants | D: Placebo Then Chloroquine for On-ART Participants
Number analyzed (Participants) | 15 | 16 | 17 | 19
percent of CD4 expressing HLA-DR+/CD38+ | 8.5 [5.5 to 12.0] | 9.8 [8.8 to 14.3] | 8.7 [6.9 to 10.0] | 9.9 [6.8 to 12.3]

16. Secondary Outcome: Percent CD4 HLA-DR+/CD38+ at Week 12
Description: Results reported are the week 12 percentage of CD4 expressing HLA-DR+/CD38+.
Time Frame: At Week 12
Population: Analysis is based on all participants with assay data at week 12.
Measure: Median (Inter-Quartile Range); unit: percent of CD4 expressing HLA-DR+/CD38+
Arm/Group | A: Chloroquine Then Placebo for Off-ART Participants | B: Placebo Then Chloroquine for Off-ART Participants | C: Chloroquine Then Placebo for On-ART Participants | D: Placebo Then Chloroquine for On-ART Participants
Number analyzed (Participants) | 14 | 16 | 16 | 19
percent of CD4 expressing HLA-DR+/CD38+ | 6.5 [4.0 to 13.0] | 10.5 [8.0 to 14.0] | 7.7 [4.2 to 9.2] | 9.0 [7.0 to 14.0]

17. Secondary Outcome: Percent CD4 HLA-DR+/CD38+ at Week 24
Description: Results reported are the week 24 percentage of CD4 expressing HLA-DR+/CD38+.
Time Frame: At Week 24
Population: Analysis is based on all participants with assay data at week 24.
Measure: Median (Inter-Quartile Range); unit: percent of CD4 expressing HLA-DR+/CD38+
Arm/Group | A: Chloroquine Then Placebo for Off-ART Participants | B: Placebo Then Chloroquine for Off-ART Participants | C: Chloroquine Then Placebo for On-ART Participants | D: Placebo Then Chloroquine for On-ART Participants
Number analyzed (Participants) | 13 | 14 | 16 | 19
percent of CD4 expressing HLA-DR+/CD38+ | 11.0 [6.0 to 14.0] | 12.5 [8.0 to 18.0] | 7.3 [6.0 to 8.5] | 9.2 [7.8 to 13.4]

18. Secondary Outcome: IL-6, Soluble TNF-rI (sTNF-rI) and D-dimer at Baseline
Description: Baseline IL-6, sTNF-rI and D-dimer were computed as the mean of pre-entry and entry IL-6, sTNF-rI and D-dimer, respectively.
Time Frame: At pre-entry and entry
Population: Analysis is based on all participants with assay data at pre-entry or entry.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | A: Chloroquine Then Placebo for Off-ART Participants | B: Placebo Then Chloroquine for Off-ART Participants | C: Chloroquine Then Placebo for On-ART Participants | D: Placebo Then Chloroquine for On-ART Participants
Number analyzed (Participants) | 15 | 16 | 17 | 19
pg/mL
  IL-6 | 1.65 [0.77 to 2.66] | 1.62 [0.97 to 1.97] | 1.01 [0.72 to 1.56] | 1.51 [1.01 to 1.92]
  sTNF-rI | 1228.66 [992.52 to 1359.06] | 1377.81 [1086.72 to 1558.35] | 1316.63 [1127.96 to 1487.45] | 1250.85 [995.60 to 1591.80]
  D-dimer | 286390 [162780 to 541950] | 328460 [188690 to 422650] | 107890 [88440 to 151810] | 103530 [71420 to 193330]

19. Secondary Outcome: IL-6, Soluble TNF-rI (sTNF-rI) and D-dimer at Week 12
Description: Results reported are the week 12 IL-6, sTNF-rI and D-dimer.
Time Frame: At week 12
Population: Analysis is based on all participants with assay data at week 12.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | A: Chloroquine Then Placebo for Off-ART Participants | B: Placebo Then Chloroquine for Off-ART Participants | C: Chloroquine Then Placebo for On-ART Participants | D: Placebo Then Chloroquine for On-ART Participants
Number analyzed (Participants) | 13 | 16 | 15 | 18
pg/mL
  IL-6 | 1.68 [0.96 to 2.35] | 1.28 [0.96 to 2.79] | 1.15 [0.79 to 2.07] | 1.30 [1.06 to 2.31]
  sTNF-rI | 1209.50 [1027.01 to 1385.70] | 1347.06 [1242.37 to 1538.05] | 1441.35 [1149.16 to 1711.86] | 1304.77 [1092.70 to 1473.54]
  D-dimer | 251320 [161660 to 621030] | 319770 [189170 to 582040] | 126540 [102190 to 179220] | 117890 [73540 to 207890]

20. Secondary Outcome: IL-6, Soluble TNF-rI (sTNF-rI) and D-dimer at Week 24
Description: Results reported are the week 24 IL-6, sTNF-rI and D-dimer.
Time Frame: At week 24
Population: Analysis is based on all participants with assay data at week 24.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | A: Chloroquine Then Placebo for Off-ART Participants | B: Placebo Then Chloroquine for Off-ART Participants | C: Chloroquine Then Placebo for On-ART Participants | D: Placebo Then Chloroquine for On-ART Participants
Number analyzed (Participants) | 14 | 16 | 16 | 19
pg/mL
  IL-6 | 1.34 [1.10 to 2.34] | 1.18 [0.84 to 2.74] | 1.02 [0.80 to 1.45] | 1.27 [1.01 to 2.33]
  sTNF-rI | 1327.21 [1056.79 to 1602.16] | 1420.30 [1229.57 to 1600.32] | 1230.21 [1063.46 to 1358.30] | 1176.20 [1060.28 to 1629.53]
  D-dimer | 264240 [210110 to 380880] | 294780 [215400 to 615550] | 100860 [78400 to 128350] | 124920 [83130 to 182450]

21. Secondary Outcome: Soluble CD14 (sCD14) at Baseline
Description: Baseline sCD14 was computed as the mean of pre-entry and entry sCD14.
Time Frame: At pre-entry and entry
Population: Analysis is based on all participants with assay data at pre-entry or entry.
Measure: Median (Inter-Quartile Range); unit: million pg/mL
Arm/Group | A: Chloroquine Then Placebo for Off-ART Participants | B: Placebo Then Chloroquine for Off-ART Participants | C: Chloroquine Then Placebo for On-ART Participants | D: Placebo Then Chloroquine for On-ART Participants
Number analyzed (Participants) | 15 | 16 | 17 | 19
million pg/mL | 1.43 [1.23 to 1.79] | 1.97 [1.77 to 2.27] | 1.80 [1.65 to 2.18] | 1.58 [1.39 to 1.87]

22. Secondary Outcome: Soluble CD14 (sCD14) at Week 12
Description: Results reported are the week 12 sCD14.
Time Frame: At week 12
Population: Analysis is based on all participants with assay data at week 12.
Measure: Median (Inter-Quartile Range); unit: million pg/mL
Arm/Group | A: Chloroquine Then Placebo for Off-ART Participants | B: Placebo Then Chloroquine for Off-ART Participants | C: Chloroquine Then Placebo for On-ART Participants | D: Placebo Then Chloroquine for On-ART Participants
Number analyzed (Participants) | 13 | 16 | 15 | 18
million pg/mL | 1.53 [1.39 to 2.05] | 1.88 [1.64 to 2.30] | 2.04 [1.60 to 2.21] | 1.63 [1.35 to 1.82]

23. Secondary Outcome: Soluble CD14 (sCD14) at Week 24
Description: Results reported are the week 24 sCD14.
Time Frame: At week 24
Population: Analysis is based on all participants with assay data at week 24.
Measure: Median (Inter-Quartile Range); unit: million pg/mL
Arm/Group | A: Chloroquine Then Placebo for Off-ART Participants | B: Placebo Then Chloroquine for Off-ART Participants | C: Chloroquine Then Placebo for On-ART Participants | D: Placebo Then Chloroquine for On-ART Participants
Number analyzed (Participants) | 14 | 16 | 16 | 19
million pg/mL | 1.53 [1.37 to 1.97] | 2.19 [1.79 to 2.35] | 1.77 [1.49 to 2.39] | 1.72 [1.54 to 2.15]

24. Secondary Outcome: Fasting Lipopolysaccharides (LPS) at Entry
Description: Results reported are for entry fasting LPS.
Time Frame: At entry
Population: Analysis is based on all participants with assay data at entry.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | A: Chloroquine Then Placebo for Off-ART Participants | B: Placebo Then Chloroquine for Off-ART Participants | C: Chloroquine Then Placebo for On-ART Participants | D: Placebo Then Chloroquine for On-ART Participants
Number analyzed (Participants) | 15 | 16 | 17 | 19
pg/mL | 13.68 [3.79 to 31.38] | 1.64 [0.70 to 28.98] | 8.00 [6.00 to 10.00] | 7.00 [2.00 to 8.00]

25. Secondary Outcome: Fasting Lipopolysaccharides (LPS) at Week 12
Description: Results reported are the week 12 fasting LPS.
Time Frame: At week 12
Population: Analysis is based on all participants with assay data at week 12.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | A: Chloroquine Then Placebo for Off-ART Participants | B: Placebo Then Chloroquine for Off-ART Participants | C: Chloroquine Then Placebo for On-ART Participants | D: Placebo Then Chloroquine for On-ART Participants
Number analyzed (Participants) | 14 | 16 | 15 | 18
pg/mL | 14.37 [4.26 to 36.63] | 13.06 [0.70 to 36.58] | 7.00 [6.00 to 9.00] | 7.00 [4.00 to 9.00]

26. Secondary Outcome: Fasting Lipopolysaccharides (LPS) at Week 24
Description: Results reported are the week 24 fasting LPS.
Time Frame: At week 24
Population: Analysis is based on all participants with assay data at week 24.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | A: Chloroquine Then Placebo for Off-ART Participants | B: Placebo Then Chloroquine for Off-ART Participants | C: Chloroquine Then Placebo for On-ART Participants | D: Placebo Then Chloroquine for On-ART Participants
Number analyzed (Participants) | 14 | 16 | 16 | 19
pg/mL | 20.54 [7.56 to 37.80] | 2.83 [0.70 to 30.57] | 7.00 [6.00 to 9.00] | 8.00 [6.00 to 10.00]

27. Secondary Outcome: Percent Activation Levels of Plasmacytoid Dendritic Cells (pDC) and Myeloid Dendritic Cells (mDC) at Baseline
Description: Baseline percent activation levels of pDC were computed as the mean of pre-entry and entry percent activation levels of pDC. Similarly, baseline percent activation levels of mDC were computed as the mean of pre-entry and entry percent activation levels of mDC.
Time Frame: At pre-entry and entry
Population: Analysis is based on all participants with assay data at pre-entry or entry.
Measure: Median (Inter-Quartile Range); unit: percentage of cells
Arm/Group | A: Chloroquine Then Placebo for Off-ART Participants | B: Placebo Then Chloroquine for Off-ART Participants | C: Chloroquine Then Placebo for On-ART Participants | D: Placebo Then Chloroquine for On-ART Participants
Number analyzed (Participants) | 16 | 17 | 18 | 19
percentage of cells
  %pDC expressing CD80+ | 0.03 [0.00 to 0.10] | 0.03 [0.00 to 0.07] | 0.13 [0.07 to 0.18] | 0.07 [0.05 to 0.20]
  %pDC expressing CD83+ | 45.48 [28.93 to 59.40] | 36.15 [27.18 to 52.28] | 19.91 [13.98 to 26.58] | 23.65 [7.49 to 27.99]
  %pDC expressing CD86+ | 9.12 [7.01 to 10.79] | 9.35 [6.33 to 11.65] | 10.96 [5.90 to 14.04] | 12.66 [8.28 to 17.91]
  %pDC expressing PDL-1+ | 2.52 [2.00 to 6.16] | 6.13 [3.01 to 12.99] | 4.48 [2.53 to 8.36] | 6.49 [2.48 to 12.03]
  %mDC expressing CD80+ | 1.04 [0.45 to 1.49] | 0.83 [0.47 to 1.01] | 1.31 [0.73 to 1.62] | 1.17 [0.76 to 2.30]
  %mDC expressing CD83+ | 38.60 [9.51 to 55.88] | 39.94 [21.98 to 59.07] | 48.17 [35.51 to 65.88] | 26.08 [12.46 to 53.69]
  %mDC expressing CD86+ | 96.29 [94.13 to 98.55] | 97.52 [95.69 to 98.50] | 96.11 [94.31 to 98.30] | 95.38 [90.57 to 96.69]
  %mDC expressing PDL-1+ | 9.82 [6.32 to 13.54] | 16.37 [7.76 to 30.19] | 4.58 [2.71 to 7.93] | 8.28 [3.08 to 11.50]

28. Secondary Outcome: Percent Activation Levels of Plasmacytoid Dendritic Cells (pDC) and Myeloid Dendritic Cells (mDC) at Week 12
Description: Results reported are the week 12 percent activation levels of pDC and mDC.
Time Frame: At week 12
Population: Analysis is based on all participants with assay data at week 12.
Measure: Median (Inter-Quartile Range); unit: percentage of cells
Arm/Group | A: Chloroquine Then Placebo for Off-ART Participants | B: Placebo Then Chloroquine for Off-ART Participants | C: Chloroquine Then Placebo for On-ART Participants | D: Placebo Then Chloroquine for On-ART Participants
Number analyzed (Participants) | 13 | 16 | 17 | 19
percentage of cells
  %pDC expressing CD80+ | 0.00 [0.00 to 0.03] | 0.05 [0.00 to 0.15] | 0.10 [0.00 to 0.20] | 0.14 [0.00 to 0.40]
  %pDC expressing CD83+ | 51.90 [22.60 to 55.60] | 40.49 [30.35 to 47.90] | 14.70 [8.28 to 24.77] | 18.20 [8.08 to 32.30]
  %pDC expressing CD86+ | 7.66 [6.50 to 8.52] | 8.48 [5.26 to 12.22] | 13.93 [6.55 to 17.84] | 13.64 [8.63 to 18.09]
  %pDC expressing PDL-1+ | 3.74 [2.66 to 5.98] | 8.43 [3.27 to 16.53] | 7.24 [2.24 to 10.67] | 5.16 [2.80 to 12.72]
  %mDC expressing CD80+ | 0.84 [0.59 to 1.12] | 1.03 [0.68 to 1.71] | 1.47 [0.95 to 1.87] | 1.01 [0.90 to 2.28]
  %mDC expressing CD83+ | 43.51 [20.34 to 51.74] | 36.47 [27.54 to 46.41] | 47.83 [32.32 to 65.29] | 26.75 [13.60 to 51.40]
  %mDC expressing CD86+ | 97.90 [96.99 to 98.51] | 97.18 [96.30 to 98.65] | 95.40 [91.26 to 97.20] | 95.15 [87.18 to 96.38]
  %mDC expressing PDL-1+ | 15.03 [9.12 to 17.48] | 16.32 [9.49 to 36.81] | 7.10 [3.18 to 10.56] | 6.09 [2.69 to 15.81]

29. Secondary Outcome: Percent Activation Levels of Plasmacytoid Dendritic Cells (pDC) and Myeloid Dendritic Cells (mDC) at Week 24
Description: Results reported are the week 24 percent activation levels of pDC and mDC.
Time Frame: At week 24
Population: Analysis is based on all participants with assay data at week 24.
Measure: Median (Inter-Quartile Range); unit: percentage of cells
Arm/Group | A: Chloroquine Then Placebo for Off-ART Participants | B: Placebo Then Chloroquine for Off-ART Participants | C: Chloroquine Then Placebo for On-ART Participants | D: Placebo Then Chloroquine for On-ART Participants
Number analyzed (Participants) | 14 | 16 | 16 | 18
percentage of cells
  %pDC expressing CD80+ | 0.05 [0.00 to 0.08] | 0.00 [0.00 to 0.05] | 0.08 [0.03 to 0.18] | 0.16 [0.05 to 0.23]
  %pDC expressing CD83+ | 44.50 [26.60 to 60.30] | 38.96 [23.17 to 45.51] | 14.80 [7.90 to 25.62] | 17.65 [7.78 to 21.44]
  %pDC expressing CD86+ | 10.13 [7.12 to 10.73] | 7.89 [4.86 to 12.61] | 11.79 [6.81 to 20.98] | 12.88 [8.99 to 19.21]
  %pDC expressing PDL-1+ | 4.34 [1.70 to 8.08] | 7.45 [2.83 to 15.09] | 5.63 [2.53 to 10.83] | 6.52 [1.05 to 12.69]
  %mDC expressing CD80+ | 0.94 [0.36 to 1.28] | 1.12 [0.67 to 1.34] | 0.76 [0.65 to 1.38] | 1.39 [0.89 to 2.00]
  %mDC expressing CD83+ | 41.21 [25.74 to 49.61] | 33.19 [24.04 to 47.68] | 36.65 [22.35 to 52.38] | 24.14 [12.93 to 36.67]
  %mDC expressing CD86+ | 97.70 [95.80 to 99.04] | 97.05 [95.40 to 98.31] | 96.69 [92.46 to 97.89] | 92.41 [89.01 to 97.20]
  %mDC expressing PDL-1+ | 9.53 [6.31 to 18.85] | 14.84 [11.11 to 40.45] | 4.13 [2.14 to 11.82] | 7.49 [3.15 to 13.64]

ADVERSE EVENTS:
Time Frame: AEs reported from start of study treatment until study completion at 28 weeks.
Description: AE reporting followed DAIDS Reporting Level, which included AEs resulting in death, congenital anomalies, fetal losses, significant disabilities, requiring hospitalization, and AEs grade 3 and higher (where grade 1=mild, 2=moderate, 3=severe, 4=life threatening/disabling, 5=death).
Arm/Group | A: Chloroquine Then Placebo for Off-ART Participants | B: Placebo Then Chloroquine for Off-ART Participants | C: Chloroquine Then Placebo for On-ART Participants | D: Placebo Then Chloroquine for On-ART Participants
Serious Adverse Events (participants affected / at risk) | 1/16 | 1/17 | 3/18 | 1/19
Other Adverse Events (participants affected / at risk) | 10/16 | 12/17 | 10/18 | 7/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A: Chloroquine Then Placebo for Off-ART Participants (N=16) | B: Placebo Then Chloroquine for Off-ART Participants (N=17) | C: Chloroquine Then Placebo for On-ART Participants (N=18) | D: Placebo Then Chloroquine for On-ART Participants (N=19)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | A: Chloroquine Then Placebo for Off-ART Participants (N=16) | B: Placebo Then Chloroquine for Off-ART Participants (N=17) | C: Chloroquine Then Placebo for On-ART Participants (N=18) | D: Placebo Then Chloroquine for On-ART Participants (N=19)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1
Blepharitis (Eye disorders) | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0
Oculogyric crisis (Eye disorders) | 0 | 0 | 1 | 0
Retinal depigmentation (Eye disorders) | 0 | 0 | 1 | 0
Retinal pigmentation (Eye disorders) | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 1 | 0
Visual impairment (Eye disorders) | 2 | 0 | 0 | 0
Anogenital dysplasia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 1
Acute hepatitis C (Infections and infestations) | 0 | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0
Genitourinary chlamydia infection (Infections and infestations) | 0 | 1 | 0 | 0
Hepatitis C (Infections and infestations) | 0 | 1 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0 | 0
Latent syphilis (Infections and infestations) | 0 | 0 | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 1
Oropharyngeal candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Secondary syphilis (Infections and infestations) | 1 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Vulvovaginitis trichomonal (Infections and infestations) | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 3 | 1 | 0
Blood albumin abnormal (Investigations) | 1 | 2 | 0 | 0
Blood alkaline phosphatase abnormal (Investigations) | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 1 | 1 | 1
Blood cholesterol (Investigations) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0
Blood glucose abnormal (Investigations) | 2 | 2 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1 | 1
Blood phosphorus decreased (Investigations) | 0 | 0 | 1 | 0
Blood potassium decreased (Investigations) | 1 | 0 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 1 | 0
Blood sodium decreased (Investigations) | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 1 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Anorectal human papilloma virus infection (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Penile wart (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 2 | 0
Acute psychosis (Psychiatric disorders) | 0 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0
Dependence (Psychiatric disorders) | 1 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 0
Hallucination, auditory (Psychiatric disorders) | 0 | 1 | 0 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0
Paranoia (Psychiatric disorders) | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1
Scrotal varicose veins (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Poor personal hygiene (Social circumstances) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No